CLINICAL TRIAL: NCT01323582
Title: Comparison of Two Macrolides, Azithromycin and Erythromycin, for Symptomatic Treatment of Gastroparesis
Acronym: AZI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original investigator left this institution, replacement investigator retired.
Sponsor: University of Florida (Other)
Collaborators: Metabolic Solutions Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 645-2008
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Gastroparesis Treatment; Gastric Emptying; Prokinetic Agents; Macrolides; Erythromycin; Azithromycin; Erythromycin Cardiac Side-effects; Erythromycin drug interactions; AZI
MeSH Terms: conditions — Gastroparesis | interventions — Erythromycin; Erythromycin Ethylsuccinate; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- erythromycin (Active Comparator): 200mg/5ml elixir administered orally three times a day half an hour prior to meals.
  Interventions: Drug: Erythromycin
- Azithromycin (Experimental): The dose of Azithromycin was determined based on our dose response curve obtained on 10 healthy subjects who were given three different doses of Azithromycin, 50 mg, 100 mg and 133 mg and underwent breath testing to determine the gastric emptying half-time. These doses were determined based on a maximum safe dosage per day of Azithromycin of 400 mg given the medication would then be administered three times daily before meals. The appearance of the medication (azithromycin) and administration period was then identical to that of Erythromycin, i.e. 5ml elixir administered orally three times a day half an hour prior to meals. The total daily dosage of Azithromycin was determined after obtaining the dose- response analysis.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Erythromycin — 200mg/5ml elixir administered orally three times a day half an hour prior to meals.
  Other Names: Erythromycin ethylsuccinate
  Arms: erythromycin
Drug: Azithromycin — The dose of Azithromycin given was determined based on the following study on 10 healthy subjects. In random order, each of ten healthy subjects underwent OBT studies following administration of AZI, at doses of 50mg, 100mg, and 133mg. The T½ and Tlag was then compared for the three doses by a randomized block analysis using Analysis of Variance followed by Tukey's multiple comparison. Results: The T½ for each of the respective doses of AZI (50mg, 100mg, and 133mg) was 129 ± 27, 128 ± 31, and 128 ± 16 minutes (p = 0.98). This data suggested that AZI at doses of 50mg, 100mg and 133 mg have fairly similar activity in its effects on gastric emptying in healthy subjects. Based on this analysis , we decided to use a dose of 50 mg/5 ml for administered TID prior to meals.
  Arms: Azithromycin

SUMMARY:
Erythromycin is effectively used in the treatment of Gastroparesis (GP) patients. In susceptible patients however, it has been associated with sudden cardiac death due to prolongation of QT intervals and subsequent cardiac risks through its interaction some other drugs. Azithromycin (AZI) is a macrolide antibiotic but does not have the mentioned druf interactions , has fewer gastrointestinal side effects, and fewer risks of QT prolongation and cardiac arrhythmias. Consequently, AZI avoids drawbacks of dosing with erythromycin and may be preferred as a prokinetic agent in patients on other concomitant medications.

We hope to demonstrate the effectiveness of Azithromycin (AZI) as compared to Erythromycin in the treatment of Gastroparesis (GP), and later, form the framework for larger randomized-controlled parallel studies to investigate use of AZI for treatment of GP.

Our novel hypothesis is to determine whether AZI can be used to treat GP.

DETAILED DESCRIPTION:
Gastroparesis (GP) is a chronic gastrointestinal motility disorder resulting from delayed transit of gastric contents from the stomach into the duodenum in the absence of mechanical outlet obstruction. The symptoms of GP are variable but include early satiety, bloating, nausea, vomiting, and epigastric abdominal pain. Although the true prevalence of the disorder is unknown, symptoms suggestive of GP are present in 7-15% of the population with an estimated one-third of diabetic patients in tertiary care settings having abnormal gastric emptying studies. Yet, despite the significant healthcare and economic costs due to frequent hospitalization in these patients, treatment of GP is difficult due to the lack of available treatment options and the often potential side effects of available prokinetic agents, including cardiac side effects such as QT prolongation, sudden cardiac death, and torsade de pointes.

One such medication used for treatment of GP is erythromycin. Erythromycin has its drawbacks. Several reports of cardiac arrhythmias associated with use of either oral or intravenous (IV) Erythromycin have been reported. This finding sparked our interest in another macrolide, Azithromycin (AZI), which does not have the drug-drug interactions as seen with erythromycin and is not metabolized by the CYP3A inhibitors, therefore having fewer cardiac side effects.

In This study our primary goal is to determine whether AZI can be used to treat GP.

ELIGIBILITY:
Inclusion Criteria:

* presenting to gastroenterology motility specialty clinics at the University of Florida (UF), who meet the clinical and radiologic diagnostic criteria for diagnosis of GP

Exclusion Criteria:

* Any history of mechanical obstruction
* Gastrointestinal malignancy
* Current use of prokinetics such as cisapride, pimozide, or anticholinergic medication which cannot be discontinued 72 hrs prior to study
* Abnormal upper endoscopy with finding of erosions or ulcerations
* Helicobacter pylori infection in past 6 months
* Recent abdominal surgery < 6 months
* Cardiac history with EKG finding of QTC > 450 done on a screening test
* Detected renal or hepatic dysfunction described as a GFR <10 ml/min and ALT/AST values > 2 times the normal level in our laboratory
* Allergy to macrolide antibiotics
* Psychiatric history other than anxiety or depression
* Predominant symptoms of irritable bowel syndrome such as constipation or diarrhea
* Uncontrolled diabetes with fasting blood glucose levels > 180 mg/dL, due to effect of hyperglycemia on gastric emptying. For patients with diabetes, blood glucose levels will be recorded in a patient diary.
* Pregnant or nursing females
* Any history of myasthenia gravis
* Current use of Coumadin, lovastatin, simvastatin Nelfinavir, theophylline, digoxin, ergotamine/dihydroergotamine products, benzodiazepines, and sildenafil (this will be discontinued for the duration of the clinical trial if subject is on this medication).
* History of elevated liver function studies or CPKs.
* Pregnancy : A urine pregnancy test will be performed at the beginning of each treatment period and only subjects who are not pregnant will be enrolled for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baharak Moshiree, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Ray WA, Murray KT, Meredith S, Narasimhulu SS, Hall K, Stein CM. Oral erythromycin and the risk of sudden death from cardiac causes. N Engl J Med. 2004 Sep 9;351(11):1089-96. doi: 10.1056/NEJMoa040582. PMID 15356306
- [Background] Frank L, Kleinman L, Ganoczy D, McQuaid K, Sloan S, Eggleston A, Tougas G, Farup C. Upper gastrointestinal symptoms in North America: prevalence and relationship to healthcare utilization and quality of life. Dig Dis Sci. 2000 Apr;45(4):809-18. doi: 10.1023/a:1005468332122. PMID 10759254
- [Background] Talley NJ, Locke GR 3rd, Lahr BD, Zinsmeister AR, Tougas G, Ligozio G, Rojavin MA, Tack J. Functional dyspepsia, delayed gastric emptying, and impaired quality of life. Gut. 2006 Jul;55(7):933-9. doi: 10.1136/gut.2005.078634. Epub 2005 Dec 1. PMID 16322108
- [Background] Soykan I, Sivri B, Sarosiek I, Kiernan B, McCallum RW. Demography, clinical characteristics, psychological and abuse profiles, treatment, and long-term follow-up of patients with gastroparesis. Dig Dis Sci. 1998 Nov;43(11):2398-404. doi: 10.1023/a:1026665728213. PMID 9824125
- [Background] Wisialowski T, Crimin K, Engtrakul J, O'Donnell J, Fermini B, Fossa AA. Differentiation of arrhythmia risk of the antibacterials moxifloxacin, erythromycin, and telithromycin based on analysis of monophasic action potential duration alternans and cardiac instability. J Pharmacol Exp Ther. 2006 Jul;318(1):352-9. doi: 10.1124/jpet.106.101881. Epub 2006 Apr 13. PMID 16614168
- [Background] Milberg P, Eckardt L, Bruns HJ, Biertz J, Ramtin S, Reinsch N, Fleischer D, Kirchhof P, Fabritz L, Breithardt G, Haverkamp W. Divergent proarrhythmic potential of macrolide antibiotics despite similar QT prolongation: fast phase 3 repolarization prevents early afterdepolarizations and torsade de pointes. J Pharmacol Exp Ther. 2002 Oct;303(1):218-25. doi: 10.1124/jpet.102.037911. PMID 12235254
- [Background] Choi MG, Camilleri M, Burton DD, Zinsmeister AR, Forstrom LA, Nair KS. [13C]octanoic acid breath test for gastric emptying of solids: accuracy, reproducibility, and comparison with scintigraphy. Gastroenterology. 1997 Apr;112(4):1155-62. doi: 10.1016/s0016-5085(97)70126-4. PMID 9097998
- [Background] Ziegler D, Schadewaldt P, Pour Mirza A, Piolot R, Schommartz B, Reinhardt M, Vosberg H, Brosicke H, Gries FA. [13C]octanoic acid breath test for non-invasive assessment of gastric emptying in diabetic patients: validation and relationship to gastric symptoms and cardiovascular autonomic function. Diabetologia. 1996 Jul;39(7):823-30. doi: 10.1007/s001250050516. PMID 8817107
- [Background] Bromer MQ, Kantor SB, Wagner DA, Knight LC, Maurer AH, Parkman HP. Simultaneous measurement of gastric emptying with a simple muffin meal using [13C]octanoate breath test and scintigraphy in normal subjects and patients with dyspeptic symptoms. Dig Dis Sci. 2002 Jul;47(7):1657-63. doi: 10.1023/a:1015856211261. PMID 12141833
- [Background] Ghoos YF, Maes BD, Geypens BJ, Mys G, Hiele MI, Rutgeerts PJ, Vantrappen G. Measurement of gastric emptying rate of solids by means of a carbon-labeled octanoic acid breath test. Gastroenterology. 1993 Jun;104(6):1640-7. doi: 10.1016/0016-5085(93)90640-x. PMID 8500721
- [Background] Nyren O, Adami HO, Bates S, Bergstrom R, Gustavsson S, Loof L, Sjoden PO. Self-rating of pain in nonulcer dyspepsia. A methodological study comparing a new fixed-point scale and the visual analogue scale. J Clin Gastroenterol. 1987 Aug;9(4):408-14. PMID 3655274
- [Background] Chey WD, Shapiro B, Zawadski A, Goodman K. Gastric emptying characteristics of a novel (13)C-octanoate-labeled muffin meal. J Clin Gastroenterol. 2001 May-Jun;32(5):394-9. doi: 10.1097/00004836-200105000-00007. PMID 11319309
- [Background] Lee JS, Camilleri M, Zinsmeister A, et al. Accurate simple measurement of gastric emptying by 13C octanoic acid breath test (OBT) in diabetes. Gastroenterology 1999; 116: G4207.
- [Background] Ware JE Jr, Snow KK, Kosinski M, Gandek B. SF-36 Health Survey: Manual and Interpretation Guide. Boston, MA: The Health Institute, New England Medical Center, 1993.
- [Background] Talley NJ, Haque M, Wyeth JW, Stace NH, Tytgat GN, Stanghellini V, Holtmann G, Verlinden M, Jones M. Development of a new dyspepsia impact scale: the Nepean Dyspepsia Index. Aliment Pharmacol Ther. 1999 Feb;13(2):225-35. doi: 10.1046/j.1365-2036.1999.00445.x. PMID 10102954

RESULTS

PARTICIPANT FLOW:
Groups:
- Erythromycin First Then Azithromycin: Erythromycin is given for 4 weeks (1-4), there is a 3 week washout (5-7), then Azithromycin is given for 4 weeks (Weeks 8-11).
- Azithromycin Then Erythromycin: Azithromycin is given for 4 weeks (1-4), there is a 3 week washout (5-7), then Erythromycin is given for 4 weeks (Weeks 8-11).
Period: Weeks 1-4 (First Period)
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Started | 12 | 14
Completed | 10 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Weeks 5-7 (Washout)
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Started | 10 | 12
Completed | 10 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Weeks 8-11 (Period 2)
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: These are all subjects who were screened, randomized, and entered the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.7) | 48.5 (11.7) | 47.4 (12.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time in Minutes for 50% of the Ingested Meal to Empty the Stomach With a Standardized Breath Test: Half the of the Week 11 Value (Period 2) Less Half the of the Week 4 Value (Period 1). This Estimates the Effect Size.
Description: Patients will be given a standardized meal enriched with a labeled material and the breath samples are then collected and analyzed. The estimated time to empty 50% (t 1/2) of the accumulated contents is recorded. Because the difference is RX-B -RX A in one group and RX A -RX B in the other, the difference between these two estimates twice the effect size. Hence the Half is applied, as is standard in the two sample method for crossover studies.
Time Frame: Weeks 4 and 11 (end of periods)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Number analyzed (Participants) | 10 | 10
Minutes | -1.6 (32.3) | -5.2 (17.9)
Statistical Analysis 1: Comparison: Erythromycin First Then Azithromycin vs Azithromycin Then Erythromycin; Study planned to accrue 50 subjects, but due to difficult recruitment was not able to meet its objective; Test type: Superiority or Other; p = 0.76, t-test, 2 sided; Satterthwaite corrected t-test was used; Mean Difference (Net) = 3.6, 95% CI 2-sided [-21.5 to 28.6], Standard Error of Mean 11.7 — A positive (negative) value would suggest AZI values would tend to be larger (smaller) than EZ values

2. Primary Outcome: Gastroparesis Cardinal Symptom Index (GCSI) Score
Description: This is a Validated instrument for measuring symptom severity in patients with gastroparesis. This scoring is based on a Likert Scale from (0-5) with zero being no symptoms and five being very severe symptoms on 9 subscales, making the overall score range from 0-45. The higher the score, the more severe patient's symptoms.
  Reference for GCSI: Revicki DA, REntz AM, Dubois D, et al. Development and validation of a patient-assessed gastroparesis symptoms severity measure: the Gastroparesis Cardinal Symptom Index. Ailment Pharm Ther 2003; 18: 141:50.
  Because the difference is RX-B -RX A in one group and RX A -RX B in the other, the difference between these two estimates twice the effect size. Hence the Half is applied, as is standard in the two sample method for crossover studies.
Time Frame: Weeks 4 and 11 (end of periods)
Population: One subject did not complete this part of analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Number analyzed (Participants) | 10 | 9
units on a scale | -1.6 (5.2) | -2.9 (7.0)
Statistical Analysis 1: Comparison: Erythromycin First Then Azithromycin vs Azithromycin Then Erythromycin; Study planned to accrue 50 subjects, but due to difficult recruitment was not able to meet its objective; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; Satterthwaite Correction used; Mean Difference (Net) = 1.3, 95% CI [-4.8 to 7.5], Standard Error of Mean 2.8 — A positive (negative) value would suggest AZI values would tend to be larger (smaller) than EZ values

3. Secondary Outcome: NDI Score
Description: Nepean Dyspepsia Index (NDI) is a measure of symptom status and quality of life in functional dyspepsia. This scale is scored using each subscale (Tension, interference with daily activities), Eating/drinking, Knowledge/control, work/study) and adding up the items for each of the five subscale score (2-10). Total score range would be 10-50).
  For the NDI, a lower number is better meaning the symptom is not effecting quality of life and a higher score closer to 50 is worse meaning it is effecting patients quality of life.
  Reference: Talley NJ, Verlinden M, Jones M. Quality of life in functional dyspepsia: responsiveness of the Nepean Dyspepsia Index and developement of a new 10-iten short form. Aliment Pharmacol Ther 2001: 15: 207-216.
  Because the difference is RX-B -RX A in one group and RX A -RX B in the other, the difference between these two estimates twice the effect size. Hence the Half is applied, as is standard in the two sample method for crossover studies.
Time Frame: Weeks 4 and 11 (end of periods)
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Number analyzed (Participants) | 10 | 10
units on a scale | 1.65 (5.6) | 1.30 (4.60)
Statistical Analysis 1: Comparison: Erythromycin First Then Azithromycin vs Azithromycin Then Erythromycin; Half of the period 2 minus period 1 differences were used, since the difference between these two derived means is an unbiased estimate of the effect size; Test type: Superiority or Other; p = 0.88, t-test, 2 sided; Satterthwaite correction for unequal standard deviations was used; Median Difference (Net) = 0.35, 95% CI 2-sided [-4.58 to 5.19], Standard Error of Mean 2.30 — A positive (negative) value would suggest AZI values would tend to be larger (smaller) than EZ values

4. Secondary Outcome: TLAG (Time From Ingestion of Meal to Start of Gastric Emptying)
Description: This is defined as the time from ingestion of the meal to the beginning of the emptying process in minutes. Because the difference is RX-B -RX A in one group and RX A -RX B in the other, the difference between these two estimates twice the effect size. Hence the Half is applied, as is standard in the two sample method for crossover studies.
Time Frame: Weeks 4 and 11 (end of periods)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Erythromycin First Then Azithromycin | Azithromycin Then Erythromycin
Number analyzed (Participants) | 10 | 10
Minutes | -1.71 (16.2) | -0.22 (8.2)
Statistical Analysis 1: Comparison: Erythromycin First Then Azithromycin vs Azithromycin Then Erythromycin; Test type: Superiority or Other; p = 0.80, t-test, 2 sided; Satterthwaite Corrected t-test; Mean Difference (Net) = -1.49, 95% CI 2-sided [-13.9 to 10.9], Standard Error of Mean 5.7 — A positive (negative) value would suggest AZI values would tend to be larger (smaller) than EZ values

5. Secondary Outcome: Change in Time to 50% Gastric Emptying: Post Test Less Baseline Pooled Over Orderings
Description: Patients will be given a standardized meal enriched with a labeled material and the breath samples are then collected and analyzed. The estimated time to reaching 50% of the accumulated contents is recorded.
Time Frame: Baseline and end of treatment period
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Erythromycin
Number analyzed (Participants) | 20
Minutes | -11.8 (40.8)
Statistical Analysis 1: Comparison: Erythromycin; Test type: Superiority or Other; p = 0.21, t-test, 2 sided; Mean Difference (Net) = -11.8, 95% CI 2-sided [-30.9 to 7.3], Standard Error of Mean 9.1 — Negative values suggest shorter emptying time post-treatment

6. Secondary Outcome: Change in Time to 50% Emptying: Post Test Less Baseline Pooled Over Orderings
Description: as for outcome 5
Time Frame: at baseline before initiation of the treatment and after completion of each treatment period.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Azithromycin: The dose of Azithromycin given was previously determined based on our dose-response analysis in 10 healthy subjects to be 50 mg. The total daily dosage of Azithromycin given therefore was 150 mg which was divided three times daily and administered as 50mg/5ml given three times a day as elixir orally, similar to the erythromycin volume.
Arm/Group | Azithromycin
Number analyzed (Participants) | 22
minutes | -15.0 (31.0)
Statistical Analysis 1: Comparison: Azithromycin; Test type: Superiority or Other; p = 0.034, t-test, 2 sided; Mean Difference (Net) = -15.0, 95% CI 2-sided [-28.7 to -1.26], Standard Error of Mean 6.61 — Negative values suggest shorter emptying time post-treatment

7. Secondary Outcome: Gastroparesis Cardinal Symptom Index (GCSI) Score Change From Baseline to Post Treatment
Description: This is a Validated instrument for measuring symptom severity in patients with gastroparesis. This scoring is based on a Likert Scale from (0-5) with zero being no symptom and five being very severe symptoms on 9 subscales, making the overall score range from 0-45. The higher the score, the more severe patient's symptoms are. The scale is reported in the references. The change was calculated by measuring the end of treatment minus baseline GCSI score.
  Negative value reflects this change.
Time Frame: Baseline and end of treatment period
Population: One subject did not complete this part of analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erythromycin
Number analyzed (Participants) | 19
units on a scale | -5.32 (8.64)
Statistical Analysis 1: Comparison: Erythromycin; Test type: Superiority or Other; p = 0.015, t-test, 2 sided; Mean Difference (Net) = -5.32, 95% CI 2-sided [-9.48 to -1.16], Standard Error of Mean 1.98 — Lower scores are favorable

8. Secondary Outcome: Does GCSI Score Improve (Lower) on Treatment, Pooling the AZ Patients Over Their Treatment Periods? Endpoint is Difference in Post-test Less Baseline
Description: This is a Validated instrument for measuring symptom severity in patients with gastroparesis. This scoring is based on a Likert Scale from (0-5) with zero being no symptom and five being very severe symptoms on 9 subscales, making the overall score range from 0-45. The higher the score, the more severe patient's symptoms are. The scale is reported in the references.
  This is a calculation taken with GCSI score at end of treatment minus baseline. Negative value reflects this change.
Time Frame: Baseline and end of treatment period
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Azithromycin
Number analyzed (Participants) | 22
units on a scale | -6.40 (10.30)
Statistical Analysis 1: Comparison: Azithromycin; Test type: Superiority or Other; p = 0.0083, t-test, 2 sided; Median Difference (Net) = -6.40, 95% CI 2-sided [-10.97 to -1.83], Standard Error of Mean 2.20 — Lower scores are favorable

ADVERSE EVENTS:
Arm/Group | Erythromycin | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 1/26 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erythromycin (N=26) | Azithromycin (N=26)
abdominal pain (Gastrointestinal disorders) | 1 | 3 — Worsening of pain while on the medication
nausea (Gastrointestinal disorders) | 0 | 3
vomiting (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No